CLINICAL TRIAL: NCT05272475
Title: The Acute Effects of Chamomile Intake on Blood Coagulation Tests in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Jonathon Schwartz, Clinical Assistant Professor, Stony Brook University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: IRB2022-00036
Record Dates: First submitted 2022-02-27; First posted 2022-03-09 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Coagulation Disorder
Keywords: Coagulation; Chamomile
MeSH Terms: conditions — Hemostatic Disorders; Thrombosis | interventions — Chamomile extract

STUDY DESIGN:
Intervention Model Description: Our study is a crossover trial with subjects randomized to one of two treatment sequences: (A) a single dose of chamomile extract capsule followed by a single dose of chamomile tea or (B) a single dose of chamomile tea followed by a single dose of chamomile extract capsule. The study requires two visit days where subjects will consume their assigned chamomile preparation at the research site. To minimize any carryover effects, the two visits must be at least 3 days apart, and no more than 8 weeks apart. Randomization will be computer-generated by the biostatistician using the SAS software, and implemented using REDCap software
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chamomile Tea (Experimental): Subjects will consume a single serving of chamomile tea on the visit day. The tea serving will be prepared using 3 grams of chamomile tea steeped in hot water according to the study protocol.
  Interventions: Dietary Supplement: Chamomile Tea
- Chamomile Extract Capsule (Experimental): Subjects will consume a single chamomile capsule on the visit day. Each capsule consists of 500 milligrams of a chamomile extract that has been standardized to 1.2% apigenin content.
  Interventions: Dietary Supplement: Chamomile Extract Capsule

INTERVENTIONS:
Dietary Supplement: Chamomile Tea — Chamomile tea bags consumed by subjects as described in study arms section.
  Arms: Chamomile Tea
Dietary Supplement: Chamomile Extract Capsule — Chamomile extract capsules consumed by subjects as described in "Experimental: Chamomile Extract Capsule" study arms section.
  Arms: Chamomile Extract Capsule

SUMMARY:
Chamomile may possess anticoagulant effects based on the presence of coumarin-like compounds within the flower. This randomized complete crossover study will investigate the impact of chamomile ingestion acutely on coagulation.

DETAILED DESCRIPTION:
Subjects will be enrolled into two groups in a crossover fashion upon obtaining written informed consent. The two intervention groups include (1) chamomile tea intake and (2) chamomile extract intake. Subjects will consume a single preparation of chamomile tea or extract capsule, and partake in a minimum of three days washout period between interventions. Screening assays of coagulation will be obtained immediately before the ingestion of chamomile, two hours after ingestion, and four hours after ingestion over the course of a single day.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed written consent
* Able to withhold use of other chamomile products (teas, lotions, supplements, extracts); will only use study-supplied chamomile products for duration of study
* Able to withhold intake of solid food at least 6 hours before intake of the chamomile preparation
* Able to withhold intake of clear liquids at least 2 hours before intake of the chamomile preparation

Exclusion Criteria:

* Past medical/family history of bleeding/thrombotic disorders (e.g. hemophilia, von-Willebrand disease)
* Chronic medications known to affect hemostasis (anticoagulants, antiplatelet agents, SSRIs, herbal/complementary medicine agents)
* Three or more alcoholic drinks daily
* Sedentary status/ restricted mobility
* Active smoker or quit smoking within one week of study period
* Females who are pregnant, breast-feeding, or lactating
* History of estrogen-dependent condition such as uterine fibroids, breast cancer, uterine cancer, or ovarian cancer
* Scheduled surgical procedure during study period
* Hospitalized patients
* Underweight (BMI < 18 kg/m2) or history of malnourishment
* Active symptoms of a respiratory, dermatologic, urinary, or gastrointestinal infection
* Diagnosed allergy to chamomile
* Severe allergy to ragweed
* Physical inability to consume chamomile tea according to the study dosing schedule
* Prescription usage of an anticoagulant agent such as warfarin, anti-Xa inhibitor, or other novel oral anticoagulants
* ADP antagonist use, including clopidogrel, prasugrel, and ticagrelor
* GPIIb/IIIa inhibitor use, including ticlopidine, eptifibatide
* More than weekly NSAID use (e.g. aspirin, ibuprofen, naproxen)
* Diagnosis of a bleeding-diathesis disorder
* Diagnosis of a hypercoagulable state
* History of elevated INR or other abnormal bleeding study (PT, aPTT, thrombin time, reptilase time, above the upper limit of normal for Stony Brook Hospital Reference Range) while not taking anticoagulants or herbal supplements listed below
* Active intake of the following herbal supplements at time of study enrollment that may alter baseline coagulation function including:

  * Ginger
  * Garlic
  * Gingko
  * Ginseng
  * Fish oil
  * Black Cohosh
  * Feverfew
  * Valerian
  * Coenzyme Q10
  * Goldenseal
  * St. John Wort
* Active intake of chamomile extracts or teas at time of study enrollment
* Inability to discontinue the aforementioned herbal supplements more than 14 days before enrollment into the study
* Significant fear of needles or fainting blood draws
* Actively taking cyclosporine
* Patient refusal to participate in study for the allotted study period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-05-12 (Actual)

PRIMARY OUTCOMES:
Change in Prothrombin Time | At two hours and four hours after the intervention

SECONDARY OUTCOMES:
Change in Activated Partial Thromboplastin Time | At two hours and four hours after the intervention
Change in Thrombin Time | At two hours and four hours after the intervention
Change in Reptilase Time | At two hours and four hours after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kimura R, Schwartz JA, Romeiser JL, Senzel L, Galanakis D, Halper D, Bennett-Guerrero E. The Acute Effect of Chamomile Intake on Blood Coagulation Tests in Healthy Volunteers: A Randomized Trial. J Appl Lab Med. 2024 May 2;9(3):468-476. doi: 10.1093/jalm/jfad120. PMID 38300838